CLINICAL TRIAL: NCT04156139
Title: High-flow Nasal Cannula Versus Noninvasive Positive Pressure Ventilation Therapy After Early Extubation for Patients With Chronic Obstructive Pulmonary Disease
Brief Title: HFNC vs NPPV After Early Extubation for Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Peking University Health Science Center (Other)
Responsible Party: Principal Investigator, Lixin Xie, Director of Department of Respiratory and Critical Care Medicine, Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018ZX09201013
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: COPD; Hypercapnic Respiratory Failure
Keywords: NPPV; HFNC; Weaning; COPD; PIC
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): NPPV treatment for patients will be performed for patients immediately after extubation in control group.
  Interventions: Device: HFNC; Device: NPPV
- intervention group (Experimental): HFNC treatment will be performed for patients immediately after extubation in the intervention group.
  Interventions: Device: HFNC; Device: NPPV

INTERVENTIONS:
Device: HFNC — The gas flow rate was set at 45~55 L/min. The inhaled oxygen concentration will be dynamically adjusted to maintain SpO2 ≥ 92%. The temperature will be set at 37 °C.
Device: NPPV — The PEEP is initially set as 5 cm H2O, the inspiratory pressure is 10 cm H2O, and the target tidal volume is 6-8 ml/kg.

SUMMARY:
High-flow nasal cannula oxygen therapy(HFNC) has proved no significant difference compared with noninvasive positive pressure ventilation (NPPV) in preventing postextubation respiratory failure and reintubation in patients with acute hypoxemic respiratory failure.However, the efficacy of early postextubation sequential HFNC in COPD patients with hypercapnic respiratory failure is inconclusive.

DETAILED DESCRIPTION:
The investigators conducted this prospective randomized controlled trial to explore the efficacy, safety of HFNC versus NPPV after early extubation in COPD patients with hypercapnic respiratory failure.The investigators hypothesized that the efficacy of HFNC after early extubation is non-inferior to that of NPPV.

ELIGIBILITY:
Inclusion Criteria:

* 1. COPD patients with bronchopulmonary infection 2. Patients with hypercapnia respiratory failure treated with invasive mechanical 3.14 days ≥ invasive mechanical ventilation ≥ 48 hours; 4.Reached the pulmonary infection control (PIC) window; 5.Have self-care ability with oxygen supply during stable phrase

Exclusion Criteria:

* Severe organ dysfunction;Myopathy or myasthenia gravis;Upper airway obstruction;A large amount of secretions and inability to drain;

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
reintubation | within the 7 days after extubation.
  The primary outcome is reintubation within the 7 days after extubation.

SECONDARY OUTCOMES:
Weaning failure | within the7 days after extubation
  Secondary Outcome is a composite criterion including reintubation events or all-cause deaths within the7 days after extubation

CONTACTS AND LOCATIONS:
Overall Officials: XIE Lixin, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No